CLINICAL TRIAL: NCT06140108
Title: Comparing the Effects of Empagliflozin and Metformin on Metabolic Dysfunction in Polycystic Ovary Syndrome With or Without Comorbidity or Multimorbidity
Brief Title: Empagliflozin vs Metformin on Metabolic Dysfunction in Polycystic Ovary Syndrome With or Without Comorbidity or Multimorbidity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SINA Health Education and Welfare Trust (Other)
Responsible Party: Principal Investigator, Hina Sharif, Assistant Manager, SINA Health Education and Welfare Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00002
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Ovary Syndrome; Weight Gain; HbA1c
MeSH Terms: conditions — Polycystic Ovary Syndrome; Weight Gain | interventions — empagliflozin; Metformin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin 10mg (Experimental): Each participant will receive empagliflozin 10mg daily for 6 months
  Interventions: Drug: Empagliflozin 10 MG
- Metformin 500mg (Active Comparator): Each participant will receive metformin 1000mg daily for 6 months
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Each participant will receive empagliflozin 10mg daily for 6 months.
  Other Names: EMPAA 10mg
  Arms: Empagliflozin 10mg
Drug: MetFORMIN 500 Mg Oral Tablet — Each participant will receive metformin 1000mg daily for 6 months.
  Other Names: Glucophage 500mg
  Arms: Metformin 500mg

SUMMARY:
this is open labelled randomize control trial among women with PCOS. PCOS, an endocrine condition, affects 5%-15% of premenopausal women. PCOS is characterized by atypical menstruation, ovulation difficulties, hyperandrogenemia, insulin resistance, and other metabolic abnormalities. Metformin is now an option for PCOS. The clinical reactions to metformin are limited and varied. Novel SGLT2 inhibitors treat type 2 diabetes with weight loss, insulin resistance reduction, and cardiovascular benefits. There is little evidence on SGLT2 inhibitor effectiveness in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

1. All women participants belong to the reproductive age group, i.e., 18 to 45 years will be included in the study.
2. All those women of BMI of greater than 25 kg/m2 will be included in this study
3. Women with a diagnosis of PCOS by using two (hyperandrogenism and oligo-anovulation) out of three (oligo-anovulation, hyperandrogenism and polycystic ovaries) Rotterdam criteria 2 which confirm hyperandrogenism (acne, seborrhea, hair loss on the scalp, increased body or facial hair) on clinical judgement will be included in the study
4. Those who documented and self-reported oligomenorrhea (cycle length greater than 35 days and nine or fewer periods per year) will be included. or
5. Those who report amenorrhea (absence of menses for a period of 3 months) will be inclusion criteria of the study.

6- PCO Women with or without comorbidity or Multimorbidity specifically, Hypothyroidism, Diabetes, Hypertension.

-

Exclusion Criteria:

1. Women of non-classical 21-hydroxylase deficiency, hyperprolactinemia, Cushing's disease, or androgen- secreting tumors will be streaked from participating.
2. In addition to this, Pregnancy or intent to become pregnant, breastfeeding, documented use of oral hormonal contraceptives and hormone- releasing implants, clomiphene citrate or oestrogen modulators, gonadotropin-releasing hormone (GnRH) modulators and Minoxidil will be excluded.
3. History or presence of malignant neoplasms within the last one years, pancreatitis (acute or chronic) will also be excluded from the study
4. Women with recurrent complaint of urinary tract infection (UTI)will be excluded from the study.

   -

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This study for women of reproductive age only
Enrollment: 70 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Irregular menstruations assessment | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  Assessment of Irregular menstruation measured by menstruations lasts 2 to 7 days after three months of treatment with either empagliflozin 10mg or metformin 1000mg daily.

SECONDARY OUTCOMES:
Body weight | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  assessment of change in Body weight in Kg after three months treatment with either empagliflozin 10mg or metformin 1000mg daily
Systolic Blood Pressure (SBP) | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  assessment of change in SBP in mm/Hg after three months treatment with either empagliflozin 10mg or metformin 1000mg daily
Lipid profile measured through biochemical test | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  assessment of change in Blood Pressure in mg/dL after three months treatment with either empagliflozin 10mg or metformin 1000mg daily
Hb1c test | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  assessment of change in Hb1c level in percentage after three months treatment with either empagliflozin 10mg or metformin 1000mg daily
fasting blood-glucose measured through biochemical test | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  assessment of fasting blood-glucose in mmol/L after three months treatment with either empagliflozin 10mg or metformin 1000mg daily
Diastolic Blood Pressure (DBP) | Six months treatment with either empagliflozin 10mg or metformin 1000mg daily
  assessment of change in DBP in mm/Hg after three months treatment with either empagliflozin 10mg or metformin 1000mg daily

CONTACTS AND LOCATIONS:
Overall Officials: Hina Sharif, PharmD,MSPH, Principal Investigator — SINA Health Education & Welfare Trust
Locations (1):
- SINA Yousuf Sb Goth, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharif H, Arsalan S, Rehman N, Muzammil A, Hatif F, Wasti F, Rehman S, Mohsin N, Nasir R, Omair W. Comparative effects of empagliflozin and metformin on metabolic dysfunction in polycystic ovary syndrome, a double blinded randomized control feasibility trial. BMC Womens Health. 2025 Nov 19;25(1):565. doi: 10.1186/s12905-025-04091-6. PMID 41257673